CLINICAL TRIAL: NCT00252798
Title: A Phase I Trial to Evaluate ZD1839(Iressa™) and Concurrent Chemo-Radiation in Patients With Locally Advanced Non Small Cell Lung Cancer
Brief Title: ZD1839 (Iressa™) and Concurrent Chemo-Radiation in Patients With Locally Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7913C00073; 1839IL/0073
Record Dates: First submitted 2005-11-01; First posted 2005-11-15 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Carboplatin; Paclitaxel; Radiation

INTERVENTIONS:
Drug: Gefitinib
Drug: Carboplatin
Drug: Paclitaxel
Procedure: Radiation

SUMMARY:
The primary objective of the trial is to determine the Maximum tolerated dose, if any, of the combination of daily ZD1839 250 mg with carboplatin AUC 2 and 60 Gray (Gy) irradiation and up to 45 mg/m2 paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced stage IIIA or IIIB NSCLC (without pleural effusion)
* Patients with apical tumours and supraclavicular nodes are acceptable if both can be easily encompassed in one radiation field
* Minimum life expectancy with treatment of 6 months
* WHO performance status 0-1

Exclusion Criteria:

* Patients with previous malignancies other than NSCLC
* Previous radiotherapy for NSCLC
* Previous immunotherapy or chemotherapy
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Forced expiratory volume in 1 second (FEV1) less than 1 litre (L)
* Absolute neutrophil count (ANC) less than 1.5 x 109/L or platelets less than 100 x 109/L
* Serum bilirubin greater than 1.25 times the upper limit of reference range
* ALT or AST greater than 2.5 times the ULRR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2002-07; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum tolerated dose, if any, of the combination of daily ZD1839 250 mg with carboplatin AUC 2 and 60 Gray (Gy) irradiation and up to 45 mg/m2 paclitaxel.

SECONDARY OUTCOMES:
To evaluate the activity potential of the combination of ZD1839, carboplatin, paclitaxel & radiation therapy
Estimating the objective response rate (complete response [CR] & partial response [PR]) as assessed by positron emission tomography with (18F)-labelled fluorodeoxyglucose (PET-FDG)
To estimate the objective response rate (CR and PR) as assessed by computerised tomography (CT) scan
To estimate the complete response rate (CR) as assessed by PET-FDG
To estimate progression free survival (PFS) as assessed by clinical examination, chest x-ray, CT scan ± PET-FDG
To estimate overall survival
To characterise the safety and tolerability of ZD1839 combined with concurrent carboplatin, paclitaxel and radiation
To determine the site of first failure (characterised as local-regional, distant or both)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Australia Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Australia (2):
  - Research Site, Woolloonabba, Queensland
  - Research Site, East Melbourne, Victoria